CLINICAL TRIAL: NCT00317278
Title: Effects of Massage on Immune System of Preterm Infants
Brief Title: Effects of Massage on the Immune System of Preterm Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Michael A Anderson, WAYNE STATE UNIVERSITY/SPONSORED PROGRAM ADMINISTRATION
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R21AT001872-01A2 (NIH)
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Premature Birth; Stress
Keywords: Massage; immune system; preterm infants
MeSH Terms: conditions — Premature Birth | interventions — Massage; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A,1 (Experimental): Massage therapy
  Interventions: Other: massage therapy
- A,2 (Sham Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Other: massage therapy — massage therapy to stable preterm infants
  Arms: A,1
Other: Sham — Sham (placebo) provided to the control group
  Arms: A,2

SUMMARY:
Infants in the Neonatal Intensive Care Unit (NICU) are exposed to stressful stimuli such as loud noises, bright lights, blood drawing, suctioning, and intubation, and are frequently left in isolation with minimal proper interaction. Stress has been demonstrated to exert a negative effect on the immune system. Different psychological interventions, including relaxation, have been used in efforts to reduce stress, and several of these techniques have been shown to improve cellular immunity. Massage therapy (MT) has been used to reduce stress in premature infants and has been associated with weight gain, shorter hospital stay, and improvement in mental/motor development. While MT has been shown to increase the number and function of natural killer (NK) cells in healthy adults and in adults infected with HIV, the effect of MT on the immune system of children, including premature infants, has never been investigated. The investigators hypothesize that, in premature infants, MT will enhance the immune system. One hundred and twenty stable premature infants meeting selection criteria will be randomized to massage and sham treatment groups. Immunologic evaluation will be performed on both groups at baseline, midway and at the end of therapy. Physicians, nurses, and parents will be masked. The investigators' unique and innovative study will be the largest study in this area and will provide valuable information on potential immune parameters associated with stress reduction and improved development in premature infants undergoing massage therapy.

DETAILED DESCRIPTION:
Already contained in Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Medically stable premature infants

Exclusion Criteria:

* Unstable premature infants with underlying medical condition

Ages: 28 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2005-10; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
NK cell numbers | baseline, midway and end of study

SECONDARY OUTCOMES:
Cellular immune function | baseline, midway and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Y. Ang, MD, Principal Investigator — Wayne State University/Detroit Medical Center
Locations (1):
- Detroit Medical Center/Wayne State University, Detroit, Michigan, United States